CLINICAL TRIAL: NCT01964131
Title: An Open Label, Randomised, Single Center, 2 Way Crossover Study to Assess Bioequivalence Between a Commercial HPMC Capsule of D961H 20 mg and a Pellets Based Sachet Formulation of D961H 20 mg by Pharmacodynamics (Intragastric pH) After Once-daily Repeated Oral Administration in Japanese Healthy Male Subjects
Brief Title: BE Study Between a Capsule and a Sachet Formulation of D961H by Pharmacodynamics in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D961TC00004
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Ulcer; Duodenal Ulcer; Anastomotic Ulcer; Reflux Esophagitis; Etc.
Keywords: Bioequivalence; pharmacodynamics; pharmacokinetics; safety; tolerability; D961H; Japanese
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- D961H sachet 20 mg (Experimental): Pellets contains esomeprazole 20 mg (esomeprazole magnesium trihydrate 22.3 mg) and excipient granules filled into single-use aluminium sachets
  Interventions: Drug: D961H sachet 20 mg
- D961H HPMC capsule 20 mg (Other): Pellets contains esomeprazole 20 mg (esomeprazole magnesium trihydrate 22.3 mg) in HPMC capsule
  Interventions: Drug: D961H HPMC capsule 20 mg

INTERVENTIONS:
Drug: D961H sachet 20 mg — Each subject will be randomised evenly to one of "Treatment: A-->B (Sequence 1)" or "Treatment: B-->A (Sequence 2)".
  Treatment A: D961H sachet 20 mg Treatment B: D961H HPMC capsule 20 mg
  Arms: D961H sachet 20 mg
Drug: D961H HPMC capsule 20 mg — Each subject will be randomised evenly to one of "Treatment: A-->B (Sequence 1)" or "Treatment: B-->A (Sequence 2)". Treatment A: D961H sachet 20 mg Treatment B: D961H HPMC capsule 20 mg
  Arms: D961H HPMC capsule 20 mg

SUMMARY:
The purpose of this study is; To investigate whether a D961H sachet 20 mg is bioequivalent to a D961H HPMC capsule 20 mg by the assessment of percentage of time with intragastric pH>4.

To compare a D961H sachet 20 mg with a D961H HPMC capsule 20 mg by the assessment of percentage of time with intragastric pH>3 during 24 hours and 24-hour median pH.

To compare PK properties of a D961H sachet 20 mg with those of D961H HPMC capsule 20 mg.

To evaluate the safety and tolerability of a D961H sachet 20 mg and D961H HPMC capsule 20 mg.

DETAILED DESCRIPTION:
The purpose of this study is; To investigate whether a pellets based sachet formulation of D961H 20 mg (D961H sachet 20 mg) is bioequivalent to a commercial HPMC capsule of D961H 20 mg (D961H HPMC capsule 20 mg) after repeated oral doses by the assessment of percentage of time with intragastric pH>4 during 24 hours after dose on Day 5.

To compare a D961H sachet 20 mg with a D961H HPMC capsule 20 mg after repeated oral doses by the assessment of percentage of time with intragastric pH>3 during 24 hours and 24-hour median pH after dose on Day 5

To compare PK properties of a D961H sachet 20 mg with those of D961H HPMC capsule 20 mg after repeated oral doses by the assessment of AUCτ, Cmax,ss, AUC0-t,ss, MRT, tmax,ss, and t1/2,ss of esomeprazole after dose on Day 5.

To evaluate the safety and tolerability of a D961H sachet 20 mg and D961H HPMC capsule 20 mg by the assessment of adverse events, clinical laboratory tests, blood pressure (BP), pulse rate and body temperature.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy Japanese male subjects between 20 and 45 years of age
* Body Mass Index (BMI=weight/height2) 19-27 (kg/m2)
* Body weight 50-85 kg
* Negative for HIV antigen/antibody, Hepatitis B surface antigen, Hepatitis C antibody and syphilis
* Clinically normal findings at the enrolment medical examination, as judged by the investigator(s)
* Homo-EM according to the genotype of CYP2C19
* Less than 30% of time with intragastric pH>4 during the baseline (pre-entry) 24-hr intragastric pH recording
* Helicobacter pylori negative has been known by urea breath test as the volunteer panel data

Exclusion Criteria:

* Significant clinical illness from the 2 weeks preceding the pre-entry visit to the randomisation, as judged by the investigator(s), eg, acute inflammatory disease which requires medical intervention
* Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease, as judged by the investigator(s), eg, sequelae of myocardial infarction, nephritis, hepatitis and cerebral infarction
* Past or present drug addiction or alcohol abuse
* Past or present severe allergic disease, hypersensitivity to food or drugs (except for seasonal hay fever), or allergic symptoms requiring medical intervention
* Moderate to heavy smoking or other sort of nicotine use (greater than 10 cigarettes per day or corresponding nicotine use)
* Clinical significant condition which could modify the absorption of the investigational product, as judged by the investigator(s), eg, effect on the absorption of the investigational product by diarrhoea, or history of excision of parts of the stomach
* Donation of blood in excess of 200 mL during the 1 month, in excess of 400 mL during the 3 months or in excess of 1200 mL during the 12 months before the first dosing of treatment period 1 (including blood component donation)
* Need for concomitant medication in the study
* Use of prescribed medication from the 2 weeks preceding the pre-entry visit to the randomisation, and over the counter (OTC) drugs (including herbs, vitamins and minerals) from one week preceding the pre-entry visit to the randomisation, unless approved by the investigator(s) and sponsor
* Use of grapefruit and grapefruit juice, and health food containing St. John's wort consumption within 2 weeks prior to the first dosing of treatment period 1
* Administration of any investigational product within 4 months preceding the pre-entry visit
* Involvement in the planning and conduct of the study (applies to all AstraZeneca staff and staff at the study site)
* Clinical judgment by the investigator(s) that the subject should not participate in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Description of whether a D961H sachet 20 mg is bioequivalent to a D961H HPMC capsule 20 mg | 27 days
  To investigate whether a D961H sachet 20 mg is bioequivalent to a D961H HPMC capsule 20 mg after repeated oral doses by the assessment of percentage of time with intragastric pH>4 during 24 hours after dose on Day 5.

SECONDARY OUTCOMES:
Description to compare a D961H sachet 20 mg with a D961H HPMC capsule 20 mg by the assessment of percentage of time with intragastric pH>3 during 24 hours and 24-hour median pH | 27 days
  To compare a D961H sachet 20 mg with a D961H HPMC capsule 20 mg after repeated oral doses by the assessment of percentage of time with intragastric pH>3 during 24 hours and 24-hour median pH after dose on Day 5
Description of the PK properties of a D961H sachet 20 mg with those of D961H HPMC capsule 20 mg. | 27 days
  To compare PK properties of a D961H sachet 20 mg with those of D961H HPMC capsule 20 mg after repeated oral doses by the assessment of AUCτ, Cmax,ss, AUC0-t,ss, MRT, tmax,ss, and t1/2,ss of esomeprazole after dose on Day 5.
Description of the safety and tolerability of a D961H sachet 20 mg and D961H HPMC capsule 20 mg. | 34 days
  To evaluate the safety and tolerability of a D961H sachet 20 mg and D961H HPMC capsule 20 mg by the assessment of adverse events, clinical laboratory tests, blood pressure (BP), pulse rate and body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Megumi Inoue, MD, PhD, Principal Investigator — Hakata Clinic Medical Co. LTA
Locations (2):
- Japan (2):
  - Hakata Clinic Medical Co. LTA, Fukuoka, Fukuoka
  - Research Site, Fukuoka, Fukuoka